CLINICAL TRIAL: NCT06790160
Title: Observational Study of Patients Being Treated With Anti-obesity Medication
Brief Title: Study of Patients Being Treated With Anti-obesity Medication
Status: Recruiting | Type: Observational
Sponsor: Texas Tech University (Other)
Collaborators: Vineyard Health Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-1109
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Obesity and Overweight
Keywords: obesity; GLP-1; body composition; nutrition; exercise
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients undergoing obesity treatment: This cohort will be comprised of individuals who are beginning obesity medication treatment at a specified virtual obesity medicine practice. Patients taking semaglutide or tirzepatide may be eligible for inclusion in this cohort.

SUMMARY:
The goal of this observational study is to learn about the real-world effects of selected obesity medications in adults undergoing medical weight management. The main outcomes of interest are changes in body composition, routine clinical markers, muscular performance, and nutritional intake over the course of treatment. Additionally, the influence of lifestyle factors on changes in these outcome variables will be examined.

Participants beginning treatment with selected obesity medications will undergo periodic body composition and muscular performance testing, as well as complete online surveys about their nutritional intake and physical activity and exercise participation. Additionally, routinely collected clinical information will be evaluated.

DETAILED DESCRIPTION:
Background. The popularity of anti-obesity medications, particularly glucagon-like peptide-1 receptor agonists (GLP-1RAs) like semaglutide and dual GLP-1/GIP receptor agonists like tirzepatide, has increased dramatically over the past several years. These medications are routinely prescribed in obesity management clinics and other medical settings. While controlled clinical trials have been conducted for specific drugs, many of these have not reported relevant outcomes, such as body composition changes, muscular performance, and nutritional intake. Additionally, these controlled clinical trials may not fully represent the "real world" effects of treatment in varied settings. As such, there is a need for observational, real-world evaluations of the effects of GLP-1RA and GLP-1/GIP drugs on body composition, muscular performance, nutritional intake, and routine clinical markers. Additionally, the influence of lifestyle factors, such as exercise participation, on the observed changes in these outcomes should be evaluated.

Overview. Eligible participants beginning treatment with selected obesity medications (semaglutide or tirzepatide) at a specified virtual health clinic will undergo periodic body composition and muscular performance testing, as well as complete online surveys about their nutritional intake and physical activity and exercise participation. Additionally, routinely collected clinical information will be evaluated.

Body Composition Assessment. Participants will be asked to report an approved local DXA testing facility for a baseline body composition assessment as close as possible to the beginning of their anti-obesity medication treatment. Participants will be requested to report for another scan after ~6 months of treatment, as well as after ~17 months of treatment (provided they are still undergoing treatment at this point).

Handgrip Strength Testing. Handgrip testing will take place using a standard, consumer-grade at-home handgrip dynamometer, which will be provided to each participant. Participants will be provided with instructions for conducting the handgrip testing. This testing will be completed at baseline (as close as possible to the initiation of anti-obesity medication), and after ~3, ~6, and ~17 months of treatment (provided they are still undergoing treatment at these time points).

Questionnaires. The following questionnaires will be completed at baseline (as close as possible to the initiation of anti-obesity medication), and after ~3, ~6, and ~17 months of treatment (provided they are still undergoing treatment at these time points):

1. Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool
2. The International Physical Activity Questionnaire (IPAQ)
3. The Muscle-Strengthening Exercise Questionnaire (MSEQ)

Standard Clinical Markers. Some clinical markers routinely collected during standard medical treatment will also be evaluated, including a lipid panel (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides), hemoglobin A1C, glucose, and blood pressure.

Power Analysis. A priori power analyses were conducted for repeated-measures ANOVA (within-subjects factors) using G*Power to determine the required sample size. The analyses used a conservative effect size (f = 0.25; "medium" strength), an alpha error probability (α) of 0.05, a desired statistical power (1-β) of 0.8, and specified one group. Ranges of number of repeated measures (2 to 4), correlations between repeated measures (0.25 to 0.5), and nonsphericity corrections (ε; 0.8 to 1) were implemented. These analyses indicated the total sample size required to achieve adequate power ranged from 24 to 50 participants. A priori power analyses were conducted for linear multiple regression (R2 deviation from zero) using G*Power to determine the required sample size for analyses examining predictors of variation in changes in outcome variables. A medium strength effect size (f2=0.15), an alpha error probability (α) of 0.05, and a desired statistical power (1-β) of 0.8 were specified. This analysis indicated that up to 6 predictors could be included in the regression model at a sample size of 98 participants. Based on consideration of these analyses, a target sample size of 100 was specified.

Statistical Analysis. Comprehensive descriptive data will be presented. Changes in all outcome variables over time will be quantified using appropriate statistical methods (e.g., repeated-measures ANOVA or a similar linear model). Additionally, the potential influence of lifestyle factors - particularly nutritional intake, physical activity level, and participation in muscle-strengthening activities - and medication type (semaglutide vs. tirzepatide) on outcome measures will be explored using an appropriate method (e.g., multiple linear regression or a related linear model, such as a linear mixed-effects model).

ELIGIBILITY:
Inclusion Criteria:

* Patient who is beginning treatment through Vineyard Virtual Health Clinic using semaglutide or tirzepatide. While the physician will individualize the treatment plans, the criteria for these medications will include, at a minimum: (A) a body mass index ≥30 kg/m2; OR (B) a BMI ≥27 kg/m2 plus at least one comorbidity.
* Patient who lives in drivable proximity to a city with an accepted DXA testing facility and is willing to report to the facility for periodic body composition testing.

Exclusion Criteria:

* Patients with type 2 diabetes.
* Patients who report not being willing or able to complete the assessments included in this research study.
* Patients who are currently pregnant or trying to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is eligible individuals who are undergoing standard obesity medication treatment at a specified virtual obesity medicine practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in Total Lean Soft Tissue | From baseline assessment to last available time point (follow-up assessments conducted ~6 months and ~17 months after baseline).
  Change in total lean soft tissue assessed by dual-energy X-ray absorptiometry.
Change in Appendicular Lean Soft Tissue | From baseline assessment to last available time point (follow-up assessments conducted ~6 months and ~17 months after baseline).
  Change in appendicular lean soft tissue assessed by dual-energy X-ray absorptiometry.
Change in Total Fat Mass | From baseline assessment to last available time point (follow-up assessments conducted ~6 months and ~17 months after baseline).
  Change in total fat mass assessed by dual-energy X-ray absorptiometry.
Change in Handgrip Strength | From baseline assessment to last available time point (follow-up assessments conducted ~3, ~6, and ~17 months after baseline).
  Change in maximal handgrip strength as determined by a handgrip dynamometer.

SECONDARY OUTCOMES:
Change in Total Body Mass | From baseline assessment to last available time point (follow-up assessments conducted ~6 months and ~17 months after baseline).
  Change in total body mass assessed by dual-energy X-ray absorptiometry.
Change in Total Body Fat Percentage | From baseline assessment to last available time point (follow-up assessments conducted ~6 months and ~17 months after baseline).
  Change in total body fat percentage assessed by dual-energy X-ray absorptiometry.
Change in Total Bone Mineral Content | From baseline assessment to last available time point (follow-up assessments conducted ~6 months and ~17 months after baseline).
  Change in total bone mineral content assessed by dual-energy X-ray absorptiometry.
Change in Visceral Fat | From baseline assessment to last available time point (follow-up assessments conducted ~6 months and ~17 months after baseline).
  Change in visceral fat assessed by dual-energy X-ray absorptiometry.

OTHER OUTCOMES:
Change in Total Cholesterol | From baseline assessment to last available time point.
  Change in total cholesterol as assessed by a lipid panel.
Change in LDL Cholesterol | From baseline assessment to last available time point.
  Change in low-density lipoprotein cholesterol as assessed by a lipid panel.
Change in HDL Cholesterol | From baseline assessment to last available time point.
  Change in high-density lipoprotein cholesterol as assessed by a lipid panel.
Change in Triglycerides | From baseline assessment to last available time point.
  Change in triglycerides as assessed by a lipid panel.
Change in Hemoglobin A1C | From baseline assessment to last available time point.
  Change in hemoglobin A1C as assessed by a routine blood panel.
Change in Glucose | From baseline assessment to last available time point.
  Change in blood glucose as assessed by a blood panel.
Change in Blood Pressure | From baseline assessment to last available time point.
  Change in blood pressure as assessed by sphygmomanometry.
Energy Intake | From baseline assessment to last available time point (follow-up assessments conducted ~3, ~6, and ~17 months after baseline).
  Total energy intake as assessed by the Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool.
Protein Intake | From baseline assessment to last available time point (follow-up assessments conducted ~3, ~6, and ~17 months after baseline).
  Total protein intake as assessed by the Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool.
Carbohydrate Intake | From baseline assessment to last available time point (follow-up assessments conducted ~3, ~6, and ~17 months after baseline).
  Total carbohydrate intake as assessed by the Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool.
Fat Intake | From baseline assessment to last available time point (follow-up assessments conducted ~3, ~6, and ~17 months after baseline).
  Total fat intake as assessed by the Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool.
Fiber Intake | From baseline assessment to last available time point (follow-up assessments conducted ~3, ~6, and ~17 months after baseline).
  Total fiber intake as assessed by the Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool.
Sugar Intake | From baseline assessment to last available time point (follow-up assessments conducted ~3, ~6, and ~17 months after baseline).
  Total sugar intake as assessed by the Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool.
Muscle-strengthening activity level | From baseline assessment to last available time point (follow-up assessments conducted ~3, ~6, and ~17 months after baseline).
  Degree of participation in muscle-strengthening activities as assessed by the Muscle-Strengthening Exercise Questionnaire (MSEQ)
Physical activity level | From baseline assessment to last available time point (follow-up assessments conducted ~3, ~6, and ~17 months after baseline).
  Physical activity level as assessed by the International Physical Activity Questionnaire (IPAQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No